CLINICAL TRIAL: NCT07342660
Title: The Therapeutic Effect of Transcranial Direct Current Stimulation and Treadmill in Children With Cerebral Palsy
Brief Title: Transcranial Direct Current Stimulation and Treadmill in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hikmat Hadoush, Dr. / Associate professor, University of Sharjah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4202019; 4322019 (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-11-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; transcranial direct current stimulation; treadmill; gait function; balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Direct Current Stimulation; Exercise Test

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS & Treadmill (Experimental): The therapeutic protocol commenced with two treadmill familiarization sessions. This was followed by ten combined treatment sessions.
  Interventions: Other: transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — The therapeutic protocol commenced with two treadmill familiarization sessions. This was followed by ten combined treatment sessions, each consisting of a 12-minute interval: a 1-minute warm-up, a 10-minute simultaneous treadmill training and tDCS therapy period, and a 1-minute cool-down. Treadmill speed was initiated at 50% of the child's maximum ground speed from the 6-Minute Walk Test (6MWT) and was progressively increased based on individual tolerance.
  Other Names: treadmill

SUMMARY:
Background: Cerebral Palsy (CP) is characterized by altered excitability in bilateral sensorimotor cortical areas. Previous research using unilateral anodal transcranial direct current stimulation (tDCS) has yielded inconsistent results, highlighting a need for alternative stimulation approaches.

Objective: This study evaluated the feasibility, safety, and preliminary efficacy of combining bilateral anodal transcranial direct current stimulation (tDCS) over the sensorimotor cortices with treadmill training in children with CP.

Methods: A within-subjects case series was conducted with five children with CP. Participants received ten sessions of treadmill training (at 50% of their maximum over-ground speed) concurrently with bilateral anodal tDCS. Outcomes, assessed pre- and post-intervention, included postural alignment (medio-lateral and anterior-posterior), ankle dorsiflexion range of motion, gait variability, walking tolerance (6-minute walk test), motor function (GMFM-66), and hip/knee range of motion. Statistical analysis was performed using paired t-tests and effect sizes (Hedges' g).

Anticipated Impact: This study will pioneer a novel bilateral tDCS montage for CP rehabilitation. The findings are expected to provide critical insights into the synergistic relationship between neuromodulation and physical training, ultimately informing more effective, evidence-based interventions to enhance motor function and participation in this population.

DETAILED DESCRIPTION:
Introduction Motor control and coordination in pediatric cerebral palsy patients have been improved through various methods. Treadmill training demonstrates efficacy in enhancing gait velocity, balance, and functional independence. Furthermore, transcranial direct current stimulation (tDCS) presents a non-invasive and safe alternative to surgical or pharmacological treatments. Collectively, these interventions have proven effective in advancing gait performance and functional capabilities in this population.

The optimal protocol for administering tDCS to pediatric cerebral palsy patients has yet to be established. Contrary to earlier studies that utilized unilateral anodal stimulation targeting the contralateral motor cortex, a hypothesis suggests that bilateral stimulation of both hemispheres could yield superior outcomes. This premise is supported by magnetoencephalography (MEG) a widespread disruption in neural excitability within both sensory-motor cortices of children with CP. This bilateral impairment occurs even in cases of unilateral lesions and contributes to reduced activation in corticospinal pathways. Accordingly, subsequent research applying unilateral anodal tDCS to the ipsilateral motor cortex (non-lesioned hemisphere) demonstrated enhancements in motor functions such as reaching skills and movement duration.

As a feasibility study, this pilot research assessed the practicality and initial effects of administering bilateral anodal tDCS concurrently with treadmill training to enhance gait parameters, range of motion, and reduce spasticity in pediatric patients with diplegic CP.

Methods Study design & participants This clinical study was approved by the IRB committee of Jordan University of Science and Technology and the King Abdullah University Hospital (#2019/420) based on the Declaration of Helsinki. Five children (aged 4-12 years) with spastic diplegic CP were enrolled. Inclusion criteria stipulated a Gross Motor Function Classification System (GMFCS) level of I-III, the ability to walk independently for at least 10 meters, and an IQ greater than 70. Key exclusion criteria included a history of orthopedic surgery, neurolytic blocks, or Botox injections in the past six months, as well as the presence of concurrent orthopedic impairments, epilepsy, intracranial metal implants, or hearing aids. In addition, voluntary written informed consent was obtained from all participant children by their legal guardians before participation in the study.

Treadmill training & tDCS intervention While prior research utilizing unilateral anodal tDCS in children with CP positioned a single anode over the C3 or C4 motor cortex and a cathode on the supra-orbital area according to the 10-20 EEG system, the present study employed a bilateral montage. Using the 10-10 EEG system for more precise placement, two anodes were positioned over the left FC1 and right FC2 regions (encompassing motor and frontal areas), with two corresponding cathodes located over the bilateral supra-orbital areas. A low current intensity of 1mA was applied.

The therapeutic protocol commenced with two treadmill familiarization sessions. This was followed by ten combined treatment sessions, each consisting of a 12-minute interval: a 1-minute warm-up, a 10-minute simultaneous treadmill training and tDCS therapy period, and a 1-minute cool-down. Treadmill speed was initiated at 50% of the child's maximum ground speed from the 6-Minute Walk Test (6MWT) and was progressively increased based on individual tolerance. Tolerance was gauged by the absence of fatigue complaints, a heart rate not exceeding 70% of maximum, and the maintenance of proper gait without shuffling. Assistants were present to provide support and verbal feedback to promote correct movement patterns.

Outcome Measures

Outcome Measures Pre- and post-intervention data were collected, including:

1. Postural alignment (medio-lateral displacement)
2. Postural alignment (anterior-posterior displacement)
3. Ankle dorsiflexion range of motion (degrees)
4. Hip range of motion (degrees)
5. Knee range of motion (degrees)
6. Walking endurance assessed using the 6-Minute Walk Test (distance in meters)
7. Gross motor function assessed using the GMFM-66 (total score)
8. Gait speed (meters/second)
9. Gait variability (dimensionless autocorrelation coefficient)

Data analysis Due to the cautions reported in the previous study of using the paired t-test with extremely small sample sizes (n = 5), the mean ± standard deviation was calculated for all outcome measures, the intervention's clinical effect size was determined using Hedges' g, with values indicating small, moderate, or large effects, and gait outcomes were measured by having each child walk a 10 m track twice before and after the intervention. Data is available.

3. Result and Discussion This study protocol is innovative in term of the tDCS stimulation protocol (bilateral anodal tDCS vs. unilateral anodal tDCS), and its outcome measures that include evaluation of the brain activity and plasticity, quantitative gait outcome measures (kinematics and kinetics), motor development, quality of life, and level of enjoyment and participation, which were not examined in one full set previously.

In addition, bilateral anodal tDCS would be feasible, and safe rehabilitation tools that would modulate the brain activity and improve the gait function, balance functions, endurance, quality of life, and level of participation and enjoyment of children with CP. Therefore, exploring such short and long-term therapeutic effects of the bilateral anodal tDCS on the children's body functions, activity and participation outcome measures provide us a promising non-invasive tool in CP rehabilitation that would be combined with many other rehabilitation tools and approaches such as behavioral therapy, virtual reality, thera suit, and many other that all used as CP rehabilitation and others neurological condition. In addition, exploring the relationship between brain activity modulation, gait functions changes, and motor development and level of participation and enjoyment would provide a better understanding of this interconnected matrix that we have to consider in our future rehabilitation approaches and strategies of children with CP, and thus serve as an important aspect that will contribute to evidence-based practice in pediatric rehabilitation Besides, it would provide us a better understanding of the mechanism behind the tDCS effects.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System (GMFCS) level of I-III
* ability to walk independently for at least 10 meters
* IQ greater than 70

Exclusion Criteria:

* history of orthopedic surgery
* history of neurolytic blocks,
* history of Botox injections in the past six months
* Presence of concurrent orthopedic impairments
* Presence of epilepsy
* Presence of intracranial metal implants

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Gait speed | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Gait speed (meters/second)
Gait variability | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Gait variability (dimensionless autocorrelation coefficient)
Walking endurance | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Walking endurance assessed using the 6-Minute Walk Test (distance in meters walked within 6 minutes intervals)
Developmental Motor function | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Gross motor function measure - Item set scale (Total Score, Higher score good motor function development, lower score poor motor function development)
Postural Alignment | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Postural alignment (medio-lateral displacement in cm)
  Postural alignment (anterior-posterior displacement in cm)

SECONDARY OUTCOMES:
Spasticity | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Modified Ashworth scale (Total Score)
Joint Range of Motion | Baseline (within 7 days prior to the first intervention session) Immediately post-intervention (within 7 days following completion of the 10-session intervention period; up to 4 weeks from baseline)
  Ankle dorsiflexion range of motion (degrees)
  Hip range of motion (degrees)
  Knee range of motion (degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Hikmat Hadoush, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the study will be made available. This will include analyzable datasets underlying the reported outcomes, such as gait parameters, range of motion measures, walking endurance (6-Minute Walk Test), and Gross Motor Function Measure (GMFM-66) scores. No direct identifiers will be shared. Supporting documentation, including the study protocol and statistical analysis plan, may also be made available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary study results and available for 5 years thereafter.
Access Criteria: De-identified IPD will be available upon reasonable request from qualified researchers for the purpose of academic, educational, or non-commercial research.